CLINICAL TRIAL: NCT06754514
Title: Boehringer Laboratories Organ Retractor Device Study
Brief Title: Organ Retractor Device Study
Status: Recruiting | Type: Observational
Sponsor: Boehringer Labs LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Retractor-01
Record Dates: First submitted 2024-10-16; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Liver Retraction During Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: liver retraction — A different way to lift the liver during bariatric surgery

SUMMARY:
This study aims to assess the safety and efficacy of an organ retraction device. The study is low risk as it is only being used in patients already undergoing primary robotic bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* undergoing minimally invasive primary bariatric surgery

Exclusion Criteria:

* known liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Identified by doctor
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Ease of use and Feasibility | During surgery
  After surgery, surgeons will be asked a series of questions and asked to rank the ease of use on a scale of 1-10

CONTACTS AND LOCATIONS:
Locations (1):
- WakeMed Health & Hospitals, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No